CLINICAL TRIAL: NCT05565703
Title: The Use of PARO to Decrease Agitation and Restlessness in Persons With Dementia and or Delirium
Brief Title: The Use of PARO to Decrease Agitation in Persons With Dementia and/or Delirium
Acronym: PARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Pamela Cacchione, Professor of Geropsychiatric Nursing, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833696
Record Dates: First submitted 2022-08-04; First posted 2022-10-04 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Dementia; Delirium
Keywords: Robotics; Nursing; nonpharmacological interventions
MeSH Terms: conditions — Dementia; Delirium

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial including an intervention and attention control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): This group is randomly selected from the Acute care for elders unit and receives a one hour intervention with the PARO robotic seal two days in a row during their hospital stay.
  Interventions: Other: PARO Robotic Seal Intervention
- Attention Control Group (Active Comparator): This group is randomly selected from the Acute Care for Elders unit and receives a one hour visit from the Researcher or research assistant two days in a row.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: PARO Robotic Seal Intervention — PARO is a therapeutic robot used to comfort PWD exhibiting agitation and restlessness (www.parorobots.com). Participants are brought out to the activity are on the ACE Unit and provided with an isolation gown to wear during their interaction with the seal. The robot is then placed on their laps for them to hold on their laps, pet, rock and pick up. The participants can also brush the robot and/or give it a bath with baby wipes. The researcher encourages participant engagement with the robot. If the participant does not want the robot on their lap it is placed on a bedside table for them to interact with.
  Arms: Intervention Group
Other: Attention Control — The participants are randomly assigned and receive a one hour visit by the researcher or research assistant
  Arms: Attention Control Group

SUMMARY:
This Clinical trial tests the efficacy of using the PARO robotic seal to decrease agitation in hospitalized older adults with dementia and/or delirium. This clinical trial also tests the efficacy of the cleaning protocol for the robot. This randomized control trial includes a one hour interaction with the PARO robot two days in a row compared to an attention control with the researcher sitting with the participant in their room for one hour two days in a row. The outcomes being evaluated include both qualitative and quantitative data. Qualitative data from videotaped interactions with the persons interacting with the PARO Robot include episodes of agitation, and emotional responses to the robot via facial expressions. The quantitative outcomes include the Agitation, use of 1:1 sitters, use of psychoactive medications and length of stay.

DETAILED DESCRIPTION:
Hospitalized persons with dementia (PWD) and or delirium superimposed on dementia (DSD) are particularly vulnerable to stress due to their decreased ability to interpret their environment and the invasive procedures required. The stress of the hospital environment can exacerbate dementia-related behaviors such as agitation and restlessness and precipitate DSD. Both can cause increased use of psychotropic medications, use of paid caregivers to provide one on one observation, costs of care, and length of stay. DSD is associated with hypoactive symptoms or hyperactive symptoms such as agitation and restlessness.

The main study outcome is agitation operationalized by the CMAI-O with restlessness operationalized by the general restlessness item on the CMAI-O defined as "fidgeting, always moving around in seat, getting up and sitting down, inability to sit still." Agitation has been associated with restless behaviors in measurement tools and consensus definitions. The International Psychogeriatric Association provided the following provisional consensus clinical and research definition of agitation in cognitive disorders "Agitation is defined broadly: 1) Occurring with patients with a cognitive impairment or dementia syndrome; 2) exhibiting behavior consistent with emotional distress; 3) manifesting in at least one of the following behaviors: excessive motor-activity (e.g. pacing, rocking, gesturing, pointing fingers, restlessness, performing repetitious mannerism); verbal aggression (e.g. yelling, speaking in an excessively loud voice, using profanity, screaming, shouting); or physical aggression (e.g. grabbing, shoving, pushing, resisting, hitting others, kicking objects or people, scratching, biting, throwing objects, hitting self, slamming doors, tearing things, and destroying property); and 4) evidencing behaviors that cause excess disability and are not solely attributable to another disorder (psychiatric, medical or substance related). In a recent concept analysis, restlessness was defined by three attributes: 1) Diffuse motor activity or motion subject to limited control judged by an observer to be excessive and/or inappropriate to the circumstances; 2) the behavior is generally non-productive or disorganized, failing to address potential underlying causes; and 3) the behavior is associated with a degree of subjective distress that is either communicated by the person with dementia or extrapolated from the behavior itself. While this is more specific than the item on the CMAI-O, the two are similar. The study protocol outlined below will be conducted on the hospital's Acute Care for the Elderly (ACE) unit. One in four admissions to the ACE unit has a diagnosis of dementia. The ACE unit has 36 beds designed to care for older adults aged ≥70 years old. ACE nurses and caregivers specialize in care of the older adult. Yet, care of the PWD with or without delirium remains challenging. Dementia or DSD-related behaviors can be difficult to console or comfort away. The ACE unit is equipped with a small activity area where PWD and persons with DSD can engage in activities. Yet, what often occurs is they are brought to this area and put in front of the television with a 1:1 caregiver sitting at their side. This rarely has a positive effect. Animal-assisted therapy (AAT) has demonstrated positive effects on agitation and restlessness in older adults. However, animals require a significant amount of care, can cause allergies, carry infections and other concerns. Due to the benefits of AAT and the recognition of its limitations, robotic animals have been introduced into clinical care. Therapeutic robotic animals have been used in the community and long-term care settings, but rarely in the acute care setting. The ACE unit is the perfect setting to pilot test the use of the therapeutic robot.

PARO (PersonAl Robot) is a relatively new therapeutic robot out of Japan currently being used in the community and long-term care settings to comfort PWD exhibiting agitation and restlessness (www.parorobots.com). PARO is used in two ways: as therapy for a predetermined purpose and a fixed time as determined by a health care provider or in unsupervised use for fun in an activity. PARO has tactile, visual, auditory, temperature, and balance sensors along with three microphones to detect sound direction and intensity. PARO recognizes its name, greetings, and a few words. PARO is equipped with a behavioral control algorithm guiding the robot's responses to the older adult's interactions. PARO has been found to reduce problematic behaviors in those with dementia in need of nursing care and lessen the burden on their families. PARO provides 1) comfort by reducing anxiety, sadness, or loneliness and relieving pain; and 2) inclusion - interaction with PARO together with caregivers and sharing fun. Eighty-five percent of persons offered the opportunity to engage with PARO had a positive therapeutic effect. PARO helps avoid the potentially dangerous side effects of antipsychotics or benzodiazepines. Most importantly, PARO has no negative side effects.

Two studies have been conducted that evaluate the use of PARO with PWD in an acute hospital setting.

Study Aims and Hypotheses

This study has 4 aims: 1) To test a standardized protocol for the introduction of PARO to PWD and persons with DSD exhibiting agitation and restlessness; 2) To evaluate the feasibility of measuring the effect of PARO on agitation and restlessness using a tablet-based assessment with the Cohen-Mansfield Agitation Inventory Observation Tool (CMAI-OT) and the Pain Assessment in Advanced Dementia (PAINAD); 3) To evaluate the feasibility of measuring the effect of PARO on the social response of PWD using The Social Interaction Tool in real-time and using videotaped interactions, and 4) To determine the effectiveness of an evidence-based cleaning protocol within and between participants.

ELIGIBILITY:
Inclusion Criteria:

* A patient on the acute Care for Elders unit
* 60 years old or older up to 110 years old
* Have a diagnosis of Alzheimer's Disease and related disorders or delirium during their current hospitalization.
* Have exhibited agitation in the hospitalization based on charge nurse report.
* Responsible party provides consent and the participant assents.
* Willing to wear an isolation gown.

Exclusion Criteria:

* On isolation
* Has excessive secretions
* Has an open wound
* Does not assent to participate

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield agitation inventory observational | Day 1 this tool is assessed at baseline
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 2 this tool is assessed at baseline
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 1 this tool is assessed again 20 minutes post baseline assessment
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 2 this tool is assessed again 20 minutes post baseline assessment
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 1 this tool is assessed 40 minutes post baseline assessment
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 2 this tool is assessed 40 minutes post baseline assessment
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 1 this tool is assessed at 60 minutes post baseline
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 2 this tool is assessed at 60 minutes post baseline
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 1 this tool is assessed at 70 minutes after the baseline
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Cohen-Mansfield agitation inventory observational | Day 2 this tool is assessed at 70 minutes after the baseline
  a 29 item observational scale for dementia and delirium related agitation behaviors- score range is 29 to 116 with higher scores indicating more agitation.
Pain in Dementia Scale | Day 1 this tool is assessed at baseline
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 2 this tool is assessed at baseline
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 1 and 2 this tool is assessed again 20 minutes post baseline assessment
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 1 this tool is assessed again 20 minutes post baseline assessment
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 2 this tool is assessed 40 minutes post baseline assessment
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 1 this tool is assessed at 60 minutes post baseline
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 2 this tool is assessed at 60 minutes post baseline
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 1 this tool is assessed at 70 minutes post the baseline
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Pain in Dementia Scale | Day 2 this tool is assessed at 70 minutes post the baseline
  This is another observational scale that identifies behaviors consistent with pain in persons with dementia. The scores range from 0 to 10 with higher scores indicating more pain.
Social Interaction Tool | Day 1 this tool is completed at the end of the 60 minute interaction with the PARO robot
  This observational tool captures the interactions between the participant and the robot during the 60 minute intervention
Social Interaction Tool | Day 2 this tool is completed at the end of the 60 minute interaction with the PARO robot
  This observational tool captures the interactions between the participant and the robot during the 60 minute intervention

SECONDARY OUTCOMES:
Number of 1:1 sitter hours | Within 6 weeks of the participant's discharge a report is reviewed online to determine the number of hours this person had a sitter while in the hospital
  Obtained for a hospital report
Number of psychoactive medications | The medications are recorded within 2 hours of the Participant's Day 1 and Day 2
  found in the electronic health record
Length of stay | Within 6 weeks of the participant's discharge the number of days are retrieved from the participant electronic records
  number of days in the hospital found in the electronic record after discharge
Emotional response to the robot | Within one year of the participants engagement with the study the videotapes are reviewed and coded.
  qualitative descriptions of the individual's response and interaction with the robot

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Z Cacchione, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen-Mansfield J. Conceptualization of agitation: results based on the Cohen-Mansfield Agitation Inventory and the Agitation Behavior Mapping Instrument. Int Psychogeriatr. 1996;8 Suppl 3:309-15; discussion 351-4. doi: 10.1017/s1041610297003530. No abstract available. PMID 9154580
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Background] Cummings J, Mintzer J, Brodaty H, Sano M, Banerjee S, Devanand DP, Gauthier S, Howard R, Lanctot K, Lyketsos CG, Peskind E, Porsteinsson AP, Reich E, Sampaio C, Steffens D, Wortmann M, Zhong K; International Psychogeriatric Association. Agitation in cognitive disorders: International Psychogeriatric Association provisional consensus clinical and research definition. Int Psychogeriatr. 2015 Jan;27(1):7-17. doi: 10.1017/S1041610214001963. Epub 2014 Oct 14. PMID 25311499
- [Background] Dodds P, Martyn K, Brown M. Infection prevention and control challenges of using a therapeutic robot. Nurs Older People. 2018 Mar 23;30(3):34-40. doi: 10.7748/nop.2018.e994. PMID 29569863
- [Background] Fick DM, Mion LC. How to try this: Delirium superimposed on dementia. Am J Nurs. 2008 Jan;108(1):52-60; quiz 61. doi: 10.1097/01.NAJ.0000304476.80530.7d. PMID 18156861
- [Background] Griffiths AW, Albertyn CP, Burnley NL, Creese B, Walwyn R, Holloway I, Safarikova J, Surr CA. Validation of the Cohen-Mansfield Agitation Inventory Observational (CMAI-O) tool. Int Psychogeriatr. 2020 Jan;32(1):75-85. doi: 10.1017/S1041610219000279. PMID 30968783
- [Background] Herr K, Bursch H, Ersek M, Miller LL, Swafford K. Use of pain-behavioral assessment tools in the nursing home: expert consensus recommendations for practice. J Gerontol Nurs. 2010 Mar;36(3):18-29; quiz 30-1. doi: 10.3928/00989134-20100108-04. PMID 20128526
- [Background] Horgas A, Miller L. Pain assessment in people with dementia. Am J Nurs. 2008 Jul;108(7):62-70; quiz 71. doi: 10.1097/01.NAJ.0000325648.01797.fc. PMID 18580131
- [Background] Moyle W, Jones CJ, Murfield JE, Thalib L, Beattie ERA, Shum DKH, O'Dwyer ST, Mervin MC, Draper BM. Use of a Robotic Seal as a Therapeutic Tool to Improve Dementia Symptoms: A Cluster-Randomized Controlled Trial. J Am Med Dir Assoc. 2017 Sep 1;18(9):766-773. doi: 10.1016/j.jamda.2017.03.018. Epub 2017 Aug 2. PMID 28780395
- [Background] Regier NG, Gitlin LN. Dementia-related restlessness: relationship to characteristics of persons with dementia and family caregivers. Int J Geriatr Psychiatry. 2018 Jan;33(1):185-192. doi: 10.1002/gps.4705. Epub 2017 Mar 23. PMID 28332736
- See also: PARO Robot Web page — https://www.parorobots.com
- See also: Living with seal robots__its sociopsychological and physiological influences on the elderly at a care house. — http://ieeexplore.ieee.org/document/4339551

DOCUMENTS (1):
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT05565703/ICF_000.pdf